CLINICAL TRIAL: NCT02890459
Title: Innovative Incentive Strategies for Sustainable HIV Testing and Antiretroviral Treatment
Brief Title: Innovative Behavioral Economics Incentives Strategies for Health
Acronym: IBIS-Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Pennsylvania (Other); Makerere University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-16876; R01MH105254 (NIH)
Record Dates: First submitted 2016-08-10; First posted 2016-09-07 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: HIV/AIDS
Keywords: HIV; incentives; behavioral economics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Aim 1 - Fixed Incentive (Active Comparator): Fixed Incentive - Prize Prize incentive - Low Prize incentive - High
  Interventions: Other: Prize incentive - Low; Other: Prize incentive - High; Behavioral: Fixed Incentive - Prize
- Aim 1 - Loss Aversion (Experimental): Loss Aversion - Prize Prize incentive - Low Prize incentive - High
  Interventions: Other: Prize incentive - Low; Other: Prize incentive - High; Behavioral: Loss Aversion - Prize
- Aim 1 - Lottery (Experimental): Lottery - Prize Prize incentive - Low Prize incentive - High
  Interventions: Other: Prize incentive - Low; Other: Prize incentive - High; Behavioral: Lottery - Prize
- Aim 2 - Standard Care (Active Comparator): Standard care Travel voucher
  Interventions: Other: Travel Voucher; Other: Standard care
- Aim 2 - Enhanced Care (Intervention) (Experimental): Escalating payment incentive Travel voucher
  Interventions: Other: Escalating payment incentive; Other: Travel Voucher; Other: Standard care
- Aim 3 Pilot - Loss Aversion (Experimental): Loss Aversion - Deposit
  Interventions: Behavioral: Loss Aversion - Deposit
- Aim 3 Pilot - Fixed Incentive (Experimental): Fixed Incentive - Voucher
  Interventions: Behavioral: Fixed Incentive - Voucher
- Aim 3 Pilot - No incentive (No Intervention): Participants will be encouraged to come for repeat HIV testing, but no incentive will be offered.
- Aim 3 Trial - Loss Aversion (Experimental): Loss Aversion - Deposit
  Interventions: Behavioral: Loss Aversion - Deposit
- Aim 3 Trial - Fixed Incentive (Experimental): Fixed Incentive - Voucher
  Interventions: Behavioral: Fixed Incentive - Voucher
- Aim 3 Trial - No incentive (No Intervention): Participants will be encouraged to come for repeat HIV testing, but no incentive will be offered.

INTERVENTIONS:
Other: Prize incentive - Low — Low expected prize value.
  Arms: Aim 1 - Fixed Incentive; Aim 1 - Loss Aversion; Aim 1 - Lottery
Other: Prize incentive - High — High expected prize value.
  Arms: Aim 1 - Fixed Incentive; Aim 1 - Loss Aversion; Aim 1 - Lottery
Other: Escalating payment incentive — The incentives will increase in value when participants are found to meet the pre-specified virologic suppression criteria at 6 weeks, 3 months and 6 months.
  If the virologic threshold for an incentive is missed at the 6 week or 3 month time-point, the subsequent incentive for an undetectable HIV viral load will be reset to the initial incentive value.
  Arms: Aim 2 - Enhanced Care (Intervention)
Other: Travel Voucher — Travel voucher to assist with linkage to care.
  Arms: Aim 2 - Enhanced Care (Intervention); Aim 2 - Standard Care
Other: Standard care — Includes HIV viral load and treatment adherence counseling.
  Arms: Aim 2 - Enhanced Care (Intervention); Aim 2 - Standard Care
Behavioral: Fixed Incentive - Prize — Men are informed that if they come for HIV testing, they will receive a specific prize (gain framing). The prize will be an item worth the same amount in US dollars as loss aversion and the expected value of a lottery prize. This gain-framed incentive resembles the form that incentives usually take in most studies and serves as a comparison to the lottery-based and loss-framed incentives.
  Arms: Aim 1 - Fixed Incentive
Behavioral: Loss Aversion - Prize — The prizes are worth approximately the same amount as the fixed incentive and expected value of a lottery prize. At the time of randomization, study staff will inform the participant that he has won a prize. Staff will ask the participant to choose a specific prize from several choices, and then provide an opportunity for the participant to see the prize. Study staff will then tell participants that they will lose the prize if they do not participate in HIV testing. In this way, the incentive is framed as a loss rather than a gain, thereby leveraging loss aversion while not requiring men in very low-income settings to experience an actual loss.
  Arms: Aim 1 - Loss Aversion
Behavioral: Lottery - Prize — Men are entered in a lottery that offers a chance to win high-value prizes after testing for HIV at a community health campaign. Staff will emphasize that only those who come for HIV testing will be entered into the lottery and that not everyone will win a prize. Participants were informed at enrollment about the list of prizes and corresponding probabilities of winning them, in terms that are understandable to men with low numeracy (e.g., "1 in 20" rather than 5%). The probabilities of winning prizes varied between 1-5%, with higher value prizes having lower probability.
  Arms: Aim 1 - Lottery
Behavioral: Fixed Incentive - Voucher — A standard gain-framed incentive arm in which participants will be offered a voucher for coming for a repeat HIV test in the future.
  Arms: Aim 3 Pilot - Fixed Incentive; Aim 3 Trial - Fixed Incentive
Behavioral: Loss Aversion - Deposit — A loss-aversion framed incentive in which participants will be asked to voluntarily make a deposit that can be retrieved, with interest on the deposit, if they come for an HIV test in the future (i.e. for repeat testing)
  Arms: Aim 3 Pilot - Loss Aversion; Aim 3 Trial - Loss Aversion

SUMMARY:
The success of combination HIV prevention efforts, including HIV treatment as prevention, hinges on universal, routine HIV testing with effective treatment after HIV diagnosis. The proposed study will evaluate the comparative effectiveness and sustainability of innovative incentive strategies, informed directly by behavioral economics and decision psychology, to promote HIV testing among men and HIV treatment among HIV-infected adults in rural Uganda.

DETAILED DESCRIPTION:
[INTRODUCTION]

The success of combination HIV prevention efforts, including HIV treatment as prevention, hinges on universal, routine HIV testing with linkage to care and antiretroviral treatment initiation after HIV diagnosis. The proposed study will evaluate the comparative effectiveness and sustainability of innovative incentive strategies, informed directly by behavioral economics and decision psychology, to promote HIV testing among men and HIV and treatment among HIV-infected adults in rural Uganda.

[OBJECTIVES]

AIM 1: Adult men living in the study communities in rural Uganda (N=3,000) will be randomized to one of three (fixed, loss aversion, and lottery) incentive approaches and different incentive amounts that encourage HIV testing. The hypothesis is that lottery and loss aversion incentives will result in significantly higher testing uptake than fixed incentives. The investigators also hypothesize that the proportion of testers in each arm who are HIV-infected (secondary outcome) will be highest with lottery-based incentives. In sub-samples of men who do and do not test, the investigators will conduct in-depth interviews to assess perceptions, attitudes and preferences related to incentives that may affect how incentives influence testing.

AIM 2: Adult men and women living in the study communities (N=400) who obtained an HIV-positive result at a community health campaign will be randomized into one of two incentive approaches that encourage HIV treatment adherence. The investigators hypothesize that a financial incentive will be more effective than no incentive in promoting HIV virologic suppression (a measure of success in ART adherence and navigation of the HIV treatment cascade) as incentives capitalize on present bias by drawing attention to a salient, immediate benefit of initiating and/or maintaining treatment, and leverage loss aversion by generating implicit loss as a result of delaying the decision to initiate ART.

AIM 3 - Pilot: In order to assess the feasibility of leveraging loss aversion to increase repeat HIV testing, HIV-negative adults who are at high risk of HIV acquisition and have just tested for HIV will be randomized into one of several different incentive strategies that encourage repeat HIV testing. The incentive arms will either: a) leverage loss-aversion by requesting participants to make an initial voluntary deposit that they will lose if they do not test for HIV at a later date; or b) use a standard gain-framed incentive strategy, in which participants are told they will receive an incentive for testing again for HIV at a later date. We will compare these two types of incentive strategies to a no incentive arm as well. Results from this pilot study will also be used to inform how best to implement loss aversion-based incentives in a larger trial, and provide preliminary data to guide sample size estimates for a larger trial comparing loss aversion vs. gain-framed incentive-based strategies vs. no incentive, on the outcome of repeat HIV testing. We hypothesize that loss aversion incentives will be feasible (i.e. ≥50% of eligible adults will be willing to participate), and will result in significantly higher testing uptake than either gain-framed incentives or no incentives.

Aim 3 - Trial. Assess the comparative effectiveness of deposit contracts (a form of incentives that leverages loss aversion) vs. gain-framed incentives, compared to no incentives (control), to promote repeat HIV testing among high-risk HIV-uninfected adults. In our Aim 3 pilot trial, we assessed the feasibility and acceptability of deposit contracts: a loss aversion-based strategy to incentivize retesting for HIV. As deposit contracts were found to be highly acceptable and feasible in our Aim 3 pilot in August-December 2017 (>90% of participants in the deposit contract group made deposits into the study contracts), we will now proceed with a larger trial of sufficient sample size to compare the effectiveness of loss aversion and gain-framed incentive approaches vs. no incentives, on the outcome of repeat HIV testing. We hypothesize that deposit contracts (loss aversion-based incentives) will result in significantly higher HIV retesting uptake 3- and 6-months after enrollment than either gain-framed incentives or no incentives.

ELIGIBILITY:
AIM 1 - TESTING TRIAL

Inclusion Criteria:

* Male
* ≥18 years
* Resident (≥6 months) in one of 4 study communities

Exclusion Criteria:

* Plan to move <6 months from study start

AIM 2 - TREATMENT TRIAL

Inclusion Criteria:

* ≥18 years
* Resident (≥6 months) in one of 4 study communities
* HIV positive

Exclusion Criteria:

* Plan to move <6 months from study start

AIM 3 - REPEAT TESTING PILOT

Inclusion Criteria:

* HIV-negative by rapid HIV antibody testing at pilot trial baseline,
* Ages 18 - 59 years old,
* Attendee of high-risk site of HIV acquisition (e.g. bars, trading centers, etc.) in the region

Exclusion Criteria:

* Intention to move away from the community in the 3 months from time of recruitment

AIM 3 - REPEAT TESTING TRIAL

Inclusion Criteria:

* HIV-negative by rapid HIV antibody testing at time of recruitment,
* Ages 18 - 59 years old,
* Reported willingness to retest for HIV in the six months following recruitment,
* Sexual risk behavior, defined as at least one of the following self-reported risks in the 12 months prior to recruitment:

  1. >1 sexual partner, or
  2. known HIV-infected sexual partner, or
  3. sexually transmitted infection, or
  4. paid or received compensation or gifts for sex.

Exclusion Criteria:

* Intention to move away from the community for >=4 consecutive months during the six months following recruitment
* A history of testing for HIV >=3 times in the 12 months prior to recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3580 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who receive an HIV test at a community health campaign between intervention groups | 6-8 weeks after enrollment; annually
  Aim 1 (IBIS HIV Testing Trial) primary outcome
Proportion of participants with HIV RNA <400 copies/mL between intervention groups | 6 months after enrollment
  Aim 2 (IBIS Treatment Trial) primary outcome
Proportion of participants randomized to loss aversion trial who make a deposit | At enrollment
  Aim 3 Pilot (IBIS Repeat HIV Testing Trial) primary outcome
Proportion of participants who complete all HIV retest visits at study venue | 6 months
  Aim 3 Trial (IBIS Repeat HIV Testing Trial) primary outcome

SECONDARY OUTCOMES:
Proportion of participants who have HIV positive result between intervention groups | 6-8 weeks after enrollment; annually
  Aim 1 (IBIS HIV Testing Trial) secondary outcome
Proportion of participants who receive an HIV test at a testing site between intervention groups | 1-3 months after enrollment
  Aim 3 Pilot (IBIS Repeat HIV Testing Trial) secondary outcome
Proportion of participants who retest for HIV at study venue at 3 months | 3-4 months after enrollment
  Aim 3 Trial (IBIS Repeat HIV Testing Trial) secondary outcome
Proportion of participants who retest for HIV at study venue at 6 months | 6-7 months after enrollment
  Aim 3 Trial (IBIS Repeat HIV Testing Trial) secondary outcome
Proportion of participants who retest for HIV at 3 months among those who made deposits | 3-4 months after enrollment
  Aim 3 Trial (IBIS Repeat HIV Testing Trial) secondary outcome
Proportion of participants who retest for HIV at 6 months among those who made deposits | 6-7 months after enrollment
  Aim 3 Trial (IBIS Repeat HIV Testing Trial) secondary outcome
Cumulative incidence of HIV seroconversion | 6-7 months after enrollment
  Aim 3 Trial (IBIS Repeat HIV Testing Trial) secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Chamie, MD, MPH, Principal Investigator — University of California, San Francisco; Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Infectious Diseases Research Collaboration, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No
N/A. Individual data may be made available upon request.

REFERENCES:
- [Result] Chamie G, Schaffer EM, Ndyabakira A, Emperador DM, Kwarisiima D, Camlin CS, Havlir DV, Kahn JG, Kamya MR, Thirumurthy H. Comparative effectiveness of novel nonmonetary incentives to promote HIV testing. AIDS. 2018 Jul 17;32(11):1443-1451. doi: 10.1097/QAD.0000000000001833. PMID 29683850
- [Result] Thirumurthy H, Ndyabakira A, Marson K, Emperador D, Kamya M, Havlir D, Kwarisiima D, Chamie G. Financial incentives for achieving and maintaining viral suppression among HIV-positive adults in Uganda: a randomised controlled trial. Lancet HIV. 2019 Mar;6(3):e155-e163. doi: 10.1016/S2352-3018(18)30330-8. Epub 2019 Jan 16. PMID 30660594
- [Result] Ndyabakira A, Chamie G, Emperador D, Marson K, Kamya MR, Havlir DV, Kwarisiima D, Thirumurthy H. Men's Beliefs About the Likelihood of Serodiscordance in Couples with an HIV-Positive Partner: Survey Evidence from Rural Uganda. AIDS Behav. 2020 Mar;24(3):967-974. doi: 10.1007/s10461-019-02531-7. PMID 31073946
- [Result] Ndyabakira A, Getahun M, Byamukama A, Emperador D, Kabageni S, Marson K, Kwarisiima D, Chamie G, Thirumurthy H, Havlir D, Kamya MR, Camlin CS. Leveraging incentives to increase HIV testing uptake among men: qualitative insights from rural Uganda. BMC Public Health. 2019 Dec 30;19(1):1763. doi: 10.1186/s12889-019-8073-6. PMID 31888589
- [Result] Schaffer EM, Gonzalez JM, Wheeler SB, Kwarisiima D, Chamie G, Thirumurthy H. Promoting HIV Testing by Men: A Discrete Choice Experiment to Elicit Preferences and Predict Uptake of Community-based Testing in Uganda. Appl Health Econ Health Policy. 2020 Jun;18(3):413-432. doi: 10.1007/s40258-019-00549-5. PMID 31981135
- [Result] Chamie G, Ndyabakira A, Marson KG, Emperador DM, Kamya MR, Havlir DV, Kwarisiima D, Thirumurthy H. A pilot randomized trial of incentive strategies to promote HIV retesting in rural Uganda. PLoS One. 2020 May 29;15(5):e0233600. doi: 10.1371/journal.pone.0233600. eCollection 2020. PMID 32470089
- [Result] Kavanagh NM, Schaffer EM, Ndyabakira A, Marson K, Havlir DV, Kamya MR, Kwarisiima D, Chamie G, Thirumurthy H. Planning prompts to promote uptake of HIV services among men: a randomised trial in rural Uganda. BMJ Glob Health. 2020 Nov;5(11):e003390. doi: 10.1136/bmjgh-2020-003390. PMID 33257417
- [Result] Marson K, Ndyabakira A, Kwarisiima D, Camlin CS, Kamya MR, Havlir D, Thirumurthy H, Chamie G. HIV retesting and risk behaviors among high-risk, HIV-uninfected adults in Uganda. AIDS Care. 2021 May;33(5):675-681. doi: 10.1080/09540121.2020.1842319. Epub 2020 Nov 10. PMID 33172300
- [Result] Chamie G, Napierala S, Agot K, Thirumurthy H. HIV testing approaches to reach the first UNAIDS 95% target in sub-Saharan Africa. Lancet HIV. 2021 Apr;8(4):e225-e236. doi: 10.1016/S2352-3018(21)00023-0. PMID 33794183
- [Result] Chamie G, Kwarisiima D, Ndyabakira A, Marson K, Camlin CS, Havlir DV, Kamya MR, Thirumurthy H. Financial incentives and deposit contracts to promote HIV retesting in Uganda: A randomized trial. PLoS Med. 2021 May 4;18(5):e1003630. doi: 10.1371/journal.pmed.1003630. eCollection 2021 May. PMID 33945526
- [Derived] Camlin CS, Marson K, Ndyabakira A, Getahun M, Emperador D, Byamukama A, Kwarisiima D, Thirumurthy H, Chamie G. Understanding the role of incentives for achieving and sustaining viral suppression: A qualitative sub-study of a financial incentives trial in Uganda. PLoS One. 2022 Jun 24;17(6):e0270180. doi: 10.1371/journal.pone.0270180. eCollection 2022. PMID 35749510